CLINICAL TRIAL: NCT07384221
Title: Clinical Investigation of the Relationship Between Disease Severity and Periodontal Status in Patients With Pemphigus Vulgaris
Brief Title: Periodontal Status and Disease Severity in Pemphigus Vulgaris Patients
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, NURIYE ISIL SAYGUN, Professor, Department of Periodontology, Saglik Bilimleri Universitesi
Other Study IDs: 2025-161
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pemphigus Vulgaris (PV); Periodontal Diseases
Keywords: Pemphigus Vulgaris; Periodontitis; Desmoglein; ODSS (Oral Disease Severity Score)
MeSH Terms: conditions — Pemphigus; Periodontal Diseases; Periodontitis | interventions — Diagnosis, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pemphigus Vulgaris Group: A comprehensive oral examination including ODSS scoring and periodontal measurements (PPD, CAL, PI, GI). Additionally, serum Desmoglein 1 and 3 levels will be retrieved from the patients' medical records for biochemical correlation.
  Interventions: Other: Clinical Periodontal and Oral Evaluation

INTERVENTIONS:
Other: Clinical Periodontal and Oral Evaluation — "Participants will undergo a comprehensive oral examination. The severity of oral mucosal involvement will be recorded using the Oral Disease Severity Score (ODSS). Clinical periodontal parameters, including Probing Pocket Depth (PPD) and Clinical Attachment Level (CAL), will be measured at six sites per tooth using a periodontal probe. Additionally, current serum Desmoglein 1 and 3 levels will be retrieved from the patients' medical records for clinical correlation."

SUMMARY:
The aim of this study is to evaluate the relationship between the severity of Pemphigus Vulgaris (a chronic autoimmune skin disease) and periodontal (gum) health. Researchers will assess disease activity using the Oral Disease Severity Score (ODSS) for mouth lesions and measure serum Desmoglein 1 and 3 levels through blood tests. These findings will be compared with clinical gum measurements, such as pocket depth and attachment levels. The study intends to determine how the clinical and biochemical severity of Pemphigus Vulgaris impacts periodontal tissues and overall oral health.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Clinically and histopathologically confirmed diagnosis of Pemphigus Vulgaris.
* Presence of at least 10 natural teeth.
* Willingness to participate and signed informed consent.

Exclusion Criteria:

* Pregnancy or lactation.
* Use of systemic antibiotics or anti-inflammatory drugs within the last 3 months.
* Periodontal treatment received within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with Pemphigus Vulgaris who are receiving treatment or follow-up at the dermatology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Oral Disease Severity Score (ODSS) | Baseline
  A clinical scoring system used to assess the severity of oral mucosal involvement in patients with Pemphigus Vulgaris. It evaluates the site and extent of lesions in the oral cavity.

SECONDARY OUTCOMES:
Serum Desmoglein 1 and 3 Levels | Baseline
  Anti-desmoglein 1 and anti-desmoglein 3 autoantibody titers as recorded in the patients' medical laboratory results. Values are measured in Relative Units per milliliter (RU/mL).
Clinical Attachment Level (CAL) | Baseline
  Measurement of the distance from the cemento-enamel junction to the base of the periodontal pocket in millimeters. Higher values indicate greater attachment loss.
Probing Pocket Depth (PPD) | Baseline
  Measurement of the distance from the gingival margin to the base of the periodontal pocket in millimeters using a periodontal probe.
Plaque Index (PI) | Baseline
  An index used to assess the thickness of plaque at the gingival margin. It evaluates oral hygiene status on a scale from 0 to 3 for each tooth surface, measured according to the criteria of Silness and Löe.
Gingival Index (GI) | Baseline
  A clinical index used to assess the severity of gingival inflammation and bleeding tendency. It evaluates the color, consistency, and bleeding of the gums on a scale from 0 to 3, measured according to the criteria of Silness and Löe.

CONTACTS AND LOCATIONS:
Overall Officials: Nuriye Işıl Saygun, Professor, Principal Investigator — University of Health Sciences, Gulhane Faculty of Dentistry, Department of Periodontology
Locations (1):
- University of Health Sciences, Gulhane Faculty of Dentistry, Department of Periodontology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy and maintain confidentiality, there are no plans to share individual participant data.